CLINICAL TRIAL: NCT01423955
Title: EPO to Protect Renal Function After Cardiac Surgery. A Phase II Double Blind Randomized Controlled Study.
Brief Title: Erythropoietin (EPO) to Protect Renal Function After Cardiac Surgery
Acronym: EPRICS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-001673-70
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Kidney Failure; Renal Failure
Keywords: Erythropoietin; Erythropoetin; Cardiac surgery; Ischemia; Reperfusion; Renal function; Cystatin C; Creatinine; Safety
MeSH Terms: conditions — Renal Insufficiency; Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo arm will receive NaCl 9mg/ml with a dose of 0.2 ml/kg. The placebo dose will be prepared prior to the surgery by a independent nurse. The calculated volume will match the volume of the active durg.
  Interventions: Drug: Placebo
- Erythropoietin (Experimental): • Active substance: Erythropoietin zeta with the ATC-code: B03XA01. The drug is a Clear colorless solution for injection. The active substance will be diluted with NaCl 9mg/ml to a to a concentration of 2000 U/ml. A dose of 400U/kg will be prepared and marked before the operation. The drug will be administrated after the anesthesia induction and before the start of surgery.
  Interventions: Drug: Erythropoietin zeta

INTERVENTIONS:
Drug: Erythropoietin zeta — The active drug will be given only once after the anesthesia induction and before the start of surgery. The active drug will be diluted to 2000U/kg and given as a single dose of 400U/kg. The dose will be prepared prior to surgery by a independent nurse.
  Other Names: Active substance: Erythropoietin zeta; Drug brand name: Retacrit®; Manufacturer and Provider: Hospira; ATC-code: B03XA01
  Arms: Erythropoietin
Drug: Placebo — Placebo arm will receive NaCl 9mg/ml with a dose of 0.2 ml/kg. The placebo dose will be prepared prior to the surgery by a independent nurse. The calculated volume will match the volume of the active durg.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential of erythropoietin in reducing risk and degree of acute kidney injury after cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury is a common complication after cardiac surgery and is associated with decreased long-term survival.

Several experimental and animal studies have showed cytoprotective, preconditioning and anti-apoptotic effects of high dose erythropoietin. Clinical studies in human have also suggested that high dose erythropoietin has preconditioning effects against injury after ischemia and reperfusion on different organs in human, such as brain, heart, liver, and kidneys.

Administration of Epo in high doses in conjunction with cardiac surgery has shown to be safe with no direct side-effects.

The investigators therefore hypothesize that a preconditioning effect of erythropoietin before cardiac surgery can reduce the level of renal dysfunction after surgery in a group with preoperative renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* The patient is scheduled for non-emergent CABG surgery.
* CyC eGFR or MDRD eGFR < 60 ml/min.
* The patient has given his/her written consent to participate

Exclusion Criteria:

* The patient has an uncontrolled hypertension.
* Hypersensitivity to the active drug.
* The patient is pregnant or is a fertile woman (<50 years).
* The patient has been treated with Erythropoietin within 4 weeks prior to the surgery.
* Preoperative CyC eGFR or MDRD eGFR is < 15, or the patient is treated with dialysis.
* The patient has a known malignancy.
* The patient is planned for Off-pump CABG surgery.
* The patient is included in other ongoing clinical trial. Yes / No
* Clinically judgment by the investigator that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in plasma cystatin C measured on day 3 postoperatively. | 3 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Bjursten, M.D. Ph.D, Principal Investigator — Region Skane
Locations (1):
- Dept Thoracic Surgery, Anestesia and Intensive Care, SUS-Lund, Lund, Sweden